CLINICAL TRIAL: NCT02563613
Title: Happy Family Kitchen Movement, A Community-based Research to Enhance Family Health, Happiness and Harmony in Hong Kong: A Cluster Randomized Controlled Trial
Brief Title: Happy Family Kitchen Movement Project
Acronym: HFKM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Council of Social Service (Other)
Responsible Party: Principal Investigator, Dr. Henry C.Y. Ho, Post-doctoral Fellow, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HFKM
Record Dates: First submitted 2015-09-25; First posted 2015-09-30 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Family Health, Happiness and Harmony; Physical Health; Psychosocial Health; Family Communication; Healthy Lifestyle
Keywords: community-based intervention; family holistic health; positive psychology; physical exercise; healthy diet
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Diet, Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Physical Exercise (PE) (Experimental): Physical exercise will be promoted through the use of one of three positive psychology themes: joy, gratitude and savoring. It will comprise of a core intervention session on physical exercise, a booster session at 1 month to consolidate the knowledge and skills that they have gained, followed by a follow-up session at 3 months on healthy diet. Trained facilitators will have the relevant knowledge and skills to carry out the intervention effectively.
  Interventions: Behavioral: Physical Exercise (PE)
- Healthy Diet (HD) (Experimental): Healthy diet will be promoted through the use of one of three positive psychology themes: joy, gratitude and savoring. It will include a core intervention session on healthy diet, a booster session at 1 month to consolidate the knowledge and skills that they have gained, followed by a follow-up session at 3 months on physical exercise. Trained facilitators will have the relevant knowledge and skills to carry out the intervention effectively.
  Interventions: Behavioral: Healthy Diet (HD)
- Wait-list Control (C) (Placebo Comparator): The control group will consist of a tea gathering session at the beginning and 1 month later, followed by a follow-up session at 3 months on physical exercise or healthy diet. The tea gathering sessions will cover topics unrelated to the intervention, such as arts and crafts workshops. Trained facilitators will have the relevant knowledge and skills to carry out the intervention effectively.
  Interventions: Other: Wait-list Control (C)

INTERVENTIONS:
Behavioral: Physical Exercise (PE) — Core session: 2 hours, Booster session: 1 hour
  Arms: Physical Exercise (PE)
Behavioral: Healthy Diet (HD) — Core session: 2 hours, Booster session: 1 hour
  Arms: Healthy Diet (HD)
Other: Wait-list Control (C) — The wait-list control group will receive the intervention at 3 months.
  Arms: Wait-list Control (C)

SUMMARY:
In recent years, Hong Kong is undergoing rapid changes together with macro social and economic trends. The increasingly complex and diverse family structure is leading to a major concern in the well-being of families, including their health, happiness and harmony (3Hs). Family life and health education should be strengthened to meet the increasing needs of healthy lifestyle promotion. In light of these concerns, the Happy Family Kitchen Movement (HFKM) project, with a focus on "FAMILY Holistic Health", will be conducted at territory-wide level in Hong Kong. HFKM is a community-based research project to develop, implement and evaluate a community-based family intervention program for improving family well-being. It is expected that participants of the community-based family interventions will gain knowledge on family holistic health and in turn promote a healthy lifestyle for 3Hs.

DETAILED DESCRIPTION:
In 2011, United Nations (UN) gathered to address the prevention and control of non-communicable diseases (NCDs) worldwide. The UN, in its Political Declaration, recognized the critical importance of reducing the level of exposure to the common modifiable risk factors for NCDs, such as physical inactivity and unhealthy diet. In Hong Kong, NCDs are responsible for more than 85% of all deaths and most of these are preventable. FAMILY Project Cohort Study (2014) also found that 88.6% of Hong Kong people had inadequate vegetable and fruit intake, 70.6% had inadequate physical exercise, 26.4% were overweight and 5.4% were obese. Hong Kong, being the most westernized and developed city of China, can take a leading role in promoting and implementing the UN Political Declaration.

Families worldwide are undergoing rapid changes together with macro, social and economic trends. Demographic shifts, economic upheavals, changing societal norms and values, both immigration across national borders and migration within nations are creating new and altered structures, processes, and relationships within families. The increasingly complex and diverse family structure is leading to a major concern in the well-being of families in Hong Kong, including their health, happiness and harmony (3Hs). Family life and health education should be strengthened to meet the increasing needs of healthy lifestyle promotion. The results from the baseline findings of FAMILY Project Cohort Study (2014) revealed that only 27.9% of the participants considered themselves to be 'happy' while 15.6% of the participants were classified as 'unhappy'. Nearly one-third (30.7%) of the participants reported having experienced at least one stressful life event in the previous year due to heavier workload (10.8%), serious health problems of a family member (6.8%), worsening financial situation (6.2%), health problems (5.1%), or death of a family member (4.7%). Furthermore, more than half of the participants (52.5%) reported having some source of dyadic conflict with family members. In response to these family and health challenges, the Happy Family Kitchen Movement (HFKM) project, with a focus on "FAMILY Holistic Health", will be conducted at territory-wide level in Hong Kong.

There are now many definitions and operationally defined terms on family health. On the functional level, the terms family health, family functioning, and healthy family are often used interchangeably (Hanson & Boyd, 1996). Family health has been described as complex system, interactions, relationships and processes with the potential to enhance both well-being and the entire household's health, and routines in the family may affect family health (Denham, 1999, 2002; Yoshikawa, 2012). Despite the different perspectives in the definitions, family health should be holistically defined, encompass both wellness and illness variables and focus on the interactive, developmental, functional, psychosocial, and health processes of family experience (Anderson & Tomlinso, 1992). Hence, the HFK Movement project will focus on "FAMILY Holistic Health" which is to emphasize a more comprehensive and wide reaching aim and includes the physical, psychological and social aspects of well-being.

Over the past six years, the FAMILY project has been working on community-based projects to promote 3Hs. Since September 2010, the Happy Family Kitchen I project (HFK) was launched in Yuen Long district, with the mission to promote 3Hs by building capacity for families on positive communication. As a component of the FAMILY Project, the HFK project had demonstrated the impact to build up an effective practice model through collaboration among various project partners. HFK II was an improved version, extended and introduced to Tsuen Wan & Kwai Tsing districts in April 2012. The School of Public Health, The University of Hong Kong, collaborated with The Hong Kong Council of Social Service in the training, design and implementation, and conducted project evaluations for HFK I & II projects, which showed that the projects were well received by the family members in Yuen Long, Tsuen Wan and Kwai Tsing districts, with significantly improved 3Hs and intervention-related behaviors. Therefore, the HFKM project is developed based on the strong foundation of the HFK projects in the previous years. In view of the physical health challenges locally and globally, the new phase of FAMILY project will put more emphasis on physical health in the upcoming three years. Following the theme on FAMILY 3Hs, the new work focus is to promote family holistic health with emphasis on the interaction and integration of physical and psychosocial health.

In Hong Kong, most 'health projects' only focus on individual's physical health and usually separate physical from mental or psychosocial health. The focus of this project not only emphasizes on individuals' health but on the family's holistic health. It is aimed to help family members influence each other for healthier lifestyles. The focus on family is a new and unique concept which is an innovative, long-term and highly sustainable at the community level. With the involvement of family members, Hong Kong families can change their lifestyles and make a difference and impact on their health. A family-focused approach will be used and a holistic perspective will be adopted to design a sustainable family holistic health intervention model in the community to meet the global health challenges.

The innovative family holistic health intervention model will emphasize on the interaction and integration of physical health and psychosocial health, based on positive psychology (Seligman, 2002; Seligman, 2011; Seligman & Csikszentmihalyi, 2000), using physical exercise and healthy diet as the platform to promote finer and fitter families, which will ultimately enhance the 3Hs. Thus, the ultimate objective of the community-based project is family holistic health for 3Hs.

In practice, innovative integrated positive psychology, public health theories and minimal methods will be used to develop brief, simple and cost-effective interventions targeted at families, in collaboration with experienced NGO partners and community stakeholders. Training workshops for the promotion of family holistic health will be conducted for the facilitators of the community-based family intervention programs. Hence, a larger number of people will be able to benefit from the program which can have greater sustainability and wider dissemination as it will be easy to administer and the costs will be low. The community-based family intervention programs will be aimed at promoting a higher level of physical exercise and a healthy diet for people of all ages which will enhance family interaction, pleasure and well-being. The use of positive psychology approach can help families develop positive attitudes and stronger motivation for healthy lifestyles. By working together with family members to have more physical exercise and consume less sugar, the process will be enjoyable with quick and measurable benefits, which will ultimately enhance sustainability within the family and beyond.

The evaluations conducted will be vigorous and evidence generating with quantitative and qualitative methods and follow-ups to assess behavioral changes and improvements in the key components of family well-being. For program development, process evaluation will also be a source for data collection.

This study has two major objectives:

1. To examine the effectiveness of positive psychology and physical exercise intervention (PE) for the promotion of family health, happiness and harmony (3Hs).
2. To examine the effectiveness of positive psychology and healthy diet intervention (HD) for the promotion of family health, happiness and harmony (3Hs).

The community-based family intervention is expected to:

1. improve family health, happiness and harmony
2. promote physical and psychosocial health
3. enhance family communication
4. encourage behaviors on positive psychology, physical exercise and healthy diet

ELIGIBILITY:
Inclusion Criteria:

* Cantonese speaking
* Intact verbal and hearing abilities for interpersonal communication
* Reading and writing abilities for questionnaire completion
* Willing to participate with 1 or more family members

Exclusion Criteria:

* Participants who fail to meet the inclusion criteria

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3419 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes in family health, happiness and harmony (3Hs) from baseline to 3 months after intervention | Before core session (up to 1 week before), immediately after core session, 1 month after core session (before booster session), 3 months after core session (before follow-up session), 3 months after core session (immediately after follow-up session)
  Family 3Hs will be assessed by the family well-being scale.

SECONDARY OUTCOMES:
Changes in behaviors on positive psychology, physical exercise and healthy diet from baseline to 3 months after intervention | Before core session (up to 1 week before), 1 month after core session (before booster session), 3 months after core session (before follow-up session)
  Theme-related behaviors will be assessed by the behavioral indicator scale.
Changes in family communication from baseline to 3 months after intervention | Before core session (up to 1 week before), 1 month after core session (before booster session), 3 months after core session (before follow-up session)
  Family communication will be assessed by the family communication scale.
Changes in life satisfaction from baseline to 3 months after intervention | Before core session (up to 1 week before), 1 month after core session (before booster session), 3 months after core session (before follow-up session)
  Life satisfaction will be assessed by the satisfaction with life scale.
Changes in subjective happiness from baseline to 3 months after intervention | Before core session (up to 1 week before), immediately after core session, 1 month after core session (before booster session), 3 months after core session (before follow-up session), 3 months after core session (immediately after follow-up session)
  Subjective happiness will be assessed by the subjective happiness scale.
Changes in mental and physical health from baseline to 3 months after intervention | Before core session (up to 1 week before), 1 month after core session (before booster session), 3 months after core session (before follow-up session)
  Mental and physical health will be assessed by the SF-12v2 health survey.
Intention to change after core session | Immediately after core session
  Intention to change one's life style after receiving the core session will be assessed by an intention to change scale.
Intention to change after follow-up session | 3 months after core session (immediately after follow-up session)
  Intention to change one's life style after receiving the follow-up session will be assessed by an intention to change scale.
Satisfaction towards core session | Immediately after core session
  Satisfaction towards the core session will be assessed by a program evaluation measure.
Satisfaction towards follow-up session | 3 months after core session (Immediately after follow-up session)
  Satisfaction towards the follow-up session will be assessed by a program evaluation measure.
The process of community-based intervention program | Up to 3 months
  The process evaluation on-site observation questionnaire will be used to assess the process of the community-based intervention programs.

OTHER OUTCOMES:
Changes in physical fitness (muscle endurance) from baseline to 3 months after intervention | Before core session (up to 1 week before), 1 month after core session (before booster session), 3 months after core session (before follow-up session)
  Muscle endurance will be assessed through a simple fitness test called seated cycling.
Changes in physical fitness (balance) from baseline to 3 months after intervention | Before core session (up to 1 week before), 1 month after core session (before booster session), 3 months after core session (before follow-up session)
  Balance will be assessed through a simple fitness test called single-leg stand.

CONTACTS AND LOCATIONS:
Overall Officials: Henry C. Y. Ho, PhD, Principal Investigator — The University of Hong Kong; Tai Hing Lam, MD, Study Chair — The University of Hong Kong; Agnes YK Lai, DN, Study Director — The University of Hong Kong
Locations (1):
- The Hong Kong Council of Social Service, Wan Chai, Hong Kong, China

REFERENCES:
- [Background] Anderson KH, Tomlinson PS. The family health system as an emerging paradigmatic view for nursing. Image J Nurs Sch. 1992 Spring;24(1):57-63. doi: 10.1111/j.1547-5069.1992.tb00700.x. PMID 1541473
- [Background] Denham SA. Family routines: a structural perspective for viewing family health. ANS Adv Nurs Sci. 2002 Jun;24(4):60-74. doi: 10.1097/00012272-200206000-00010. PMID 12699277
- [Background] Denham, S. A. (1999). Part I: The definition and practice of family health. Journal of Family Nursing, 5(2), 133-159.
- [Background] Hanson, S. M., & Boyd, S. T. (1996). Family nursing: An overview. In S. M. Hanson & S. T. Boyd (Eds.), Family health care nursing: Theory, practice, and research (pp. 5-37). Philadelphia: F. A. Davis.
- [Background] Seligman, M. E. P. (2002). Authentic happiness: Using the new positive psychology to realize your potential for lasting fulfilment. New York: Free Press.
- [Background] Seligman, M. E. P. (2011). Flourish: A visionary new understanding of happiness and well-being. New York, NY: Free Press.
- [Background] Seligman ME, Csikszentmihalyi M. Positive psychology. An introduction. Am Psychol. 2000 Jan;55(1):5-14. doi: 10.1037//0003-066x.55.1.5. PMID 11392865
- [Background] The FAMILY Project. (2014). FAMILY project cohort study: Baseline findings. Hong Kong Jockey Club Charities Trust Fund and the School of Public Health, The University of Hong Kong.
- [Background] United Nations. (2011). Political declaration of the high-level meeting of the general assembly on the prevention and control of non-communicable diseases. Retrieved from http://ncdalliance.org/sites/default/files/rfiles/UN%20HLM%20Political%20Declaration%20English.pdf
- [Background] Yoshikawa H. Integrating methods in the science of family health: new directions from an institute of medicine workshop report. Arch Pediatr Adolesc Med. 2012 Jul 1;166(7):659-61. doi: 10.1001/archpediatrics.2012.510. No abstract available. PMID 22751883
- [Derived] Guo N, Ho HCY, Wang MP, Lai AY, Luk TT, Viswanath K, Chan SS, Lam TH. Factor Structure and Psychometric Properties of the Family Communication Scale in the Chinese Population. Front Psychol. 2021 Nov 12;12:736514. doi: 10.3389/fpsyg.2021.736514. eCollection 2021. PMID 34867617
- [Derived] Ho HCY, Mui MW, Wan A, Yew CW, Lam TH. A cluster randomized controlled trial of a positive physical activity intervention. Health Psychol. 2020 Aug;39(8):667-678. doi: 10.1037/hea0000885. Epub 2020 May 14. PMID 32406728